CLINICAL TRIAL: NCT03999138
Title: MRI Assessment of Pulmonary Edema in Acute Heart Failure
Acronym: MAP-AHF
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Pro00091033
Record Dates: First submitted 2019-05-22; First posted 2019-06-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acute Heart Failure; Pulmonary Edema With Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI studies (non-contrast) will consist of a free-breathing localizer (~10 seconds) followed by a free-breathing yarnball water density scan, for a total MRI time of < 3 minutes.

SUMMARY:
Researchers are testing a more accurate way to measure how much fluid is in the lungs (also called pulmonary edema, or "increased lung water") in people with Heart Failure (HF) using MRI (Magnetic Resonance Imaging). There is little known about the exact level of lung water in patients with AHF or how these levels change from the time of hospital admission to discharge. The purpose of this research study is to measure the lung water in patients hospitalized for HF, to determine the change in lung water over the course of hospitalization and treatment, and to find out if lung water levels can predict if patients are higher or lower risk for returning to the hospital or dying from heart failure.

DETAILED DESCRIPTION:
Heart failure is a condition where the heart is unable to pump enough blood to meet the body's needs and Acute Heart Failure is a sudden worsening of this condition. It is associated with many symptoms but most commonly includes shortness of breath due to pulmonary edema (or increased "lung water").

A physical exam and chest x-ray are commonly used to diagnose AHF and estimate the amount of increased lung water in patients with AHF. This study will use images from MRI (Magnetic Resonance Imaging) scans to obtain a more accurate measurement of the increased lung water in AHF patients. Lung water will be measured via MRI at hospital admission and discharge to find out the change in lung water over the course of hospitalization and treatment. The investigators will collect NT-proBNP and perform a chest x-ray upon hospital admission and again upon discharge, if not already done as part of usual care. The investigators will follow medical records for up to 5 years after hospitalization to see if the accurate lung water measurements obtained in hospital can predict long term outcomes. This is a multi-centre project and a total of 300 patients will be recruited to participate.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and willing/able to provide informed consent
* patients being treated for acute heart failure (including those patients with both reduced and preserved ejection fraction)
* patients receiving medical therapy for pulmonary edema by current standard of care (including oral or IV diuretics)
* patients identified within 48 hours of initiation of medical therapy for pulmonary edema, defined as the time of first diuretic (IV or PO) or escalation of existing diuretic therapy administered within the ED or hospital

Exclusion Criteria:

* contraindication to MRI
* patient too critically ill/unstable as per the clinical care team for transport to MRI scanner within the required scanning window
* moderate to severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with a diagnosis of acute heart failure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Magnitude of lung water density measured with MRI at Hospital Admission | Baseline (hospital admission)
  Lung water density (0-100%) is the fraction of lung tissue that contains water
Difference in lung water density measured with MRI at hospital admission and hospital discharge | 7 days
  Absolute change in lung water density from baseline (hospital admission) to hospital discharge. Lung water density will be 0%-100% at each time point.
Number and timing of clinical events and their statistical association with Outcome 1 (Magnitude of lung water density measured with MRI at Hospital Admission) | Up to 5 years
  Clinical events include cardiovascular hospitalization, cardiovascular emergency department visits or death
Number and timing of clinical events and their statistical association with Outcome 2 (Difference in lung water density measured with MRI at hospital admission and hospital discharge) | Up to 5 years
  Clinical events include cardiovascular hospitalization, cardiovascular emergency

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No